CLINICAL TRIAL: NCT01765686
Title: Randomized Controlled Trial Comparing the Utility of an Ultrasonic Coagulating Device (UCSD) With Electrothermal Bipolar Vessel Sealer (EBVS) in Thyroid Surgery.
Brief Title: Comparing Harmonic Ultrasonic Scalpel to Small Jaw Bipolar Device in Thyroid Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCCS ED 2011739D
Record Dates: First submitted 2012-12-13; First posted 2013-01-10 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Thyroid Diseases
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Harmonic (Active Comparator): Harmonic scalpel uses ultrasound technology to coagulate and to cut tissues.
  Interventions: Device: Harmonic Scalpel (Ethicon Endo-Surgery, USA)
- Small Jaw (Active Comparator): Small Jaw device uses bipolar electrical energy and pressure to form a seal and a micro blade to divide the sealed tissues.
  Interventions: Device: Ligasure Small Jaw (Covidien, USA)

INTERVENTIONS:
Device: Harmonic Scalpel (Ethicon Endo-Surgery, USA)
  Arms: Harmonic
Device: Ligasure Small Jaw (Covidien, USA)
  Arms: Small Jaw

SUMMARY:
Energy devices are used routinely during thyroid surgery to aid surgical dissection and to stop bleeding. The newer generation energy devices have several advantages over older machines. The two most commonly used newer generation energy devices are the Harmonic scalpel and the Small Jaw bipolar device. Currently there has been no randomized controlled trial that compares both devices side to side. We aim to compare the effectiveness of these two newer generation energy devices in thyroid surgery.

DETAILED DESCRIPTION:
Energy devices are used routinely during thyroid surgery to aid surgical dissection and haemostasis. The newer generation energy devices have several advantages over older machines. First, the newer devices deliver more focussed thermal application and thus are less likely to cause collateral injury to surrounding healthy tissue. This is particularly relevant in thyroid surgery because the thyroid gland is in close proximity to vital nerves that control our airway and glands that regulate calcium metabolism. Secondly, the newer energy devices have multifunctional properties and are capable of sealing, blunt dissection, grasping and dividing tissue. This is advantageous in thyroid surgery as the operating field has many narrow areas within and the potential reduction in the exchange of instruments facilitates surgery.

Currently, two of these newer generation energy devices are available for use in Singapore General Hospital and National Cancer Centre Singapore. Both devices are similarly priced; one is based on an ultrasonic vibrating blade (UCSD) to cut and coagulate tissue while the other uses bipolar electrical energy and pressure to form a seal and a micro blade to divide the sealed tissue (EBVS). To date, clinical studies comparing both devices have only been done on animal models and focus on sealing times in animal blood vessels.

We aim to compare the effectiveness of these two newer generation energy devices in thyroid surgery by looking at the incidence of post surgical complications, post operative drainage as well as the ease of use as reflected in the operating time.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-75
* Histological confirmation of differentiated thyroid cancer requiring surgery, symptomatic goiters, thyroid nodules requiring histological analysis, or thyrotoxicosis poorly controlled my medication
* Undergoing thyroid surgery

Exclusion Criteria:

* Previous neck radiotherapy
* Previous neck surgery
* Patients with advanced disease that would require radical or modified neck dissection
* Patients with lobe larger than 10 cm or nodule larger than 8 cm which requires extensive dissection that may confound the study
* Patients with connective tissue diseases or chronic diseases on long-term medications that may interfere with wound healing such as steroids.
* Patients with bleeding diatheses.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-12; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Duration of Surgery | Day 1: Day of Surgery
  Kife to skin time to closure time.
Bleeding | Day 1 and on day of drain removal.
  Measured blood loss during surgery including suction amount minus the irrigation fluid used as well as the number of gauzes. Drain amount is also recorded postoperatively

SECONDARY OUTCOMES:
Post op complications | Day 2
  Voice hoarseness, adverse events, stridor, difficulty breathing and other common complications of thyroid surgery are recorded.
Ease of use | Day 1
  Surgeon's comment on ease of use, number of nerve identified, number of parathyroid gland identified, staff's inputs on ease of use.
Vocal chords on nasal scope inspection | Day 15 and up to 3-months post-op
  Nasal scope will be done for all subjects at 2-week post operative. If normal, subject does not need to undergo the 2nd nasal scope at 3-month visit.
Ease of use | Day 1
  Measure interruption to device use, absolute failure that necessitates equipment changes, incomplete hemostasis requiring additional tying with silk sutures.

CONTACTS AND LOCATIONS:
Overall Officials: Gopal Iyer, Consultant, Principal Investigator — National Cancer Centre, Singapore; Jeremy Ng, Consultant, Principal Investigator — Singapore General Hospital; Khoon Hiang Tan, Senior Consultant, Principal Investigator — National Cancer Centre, Singapore; Chye Ngian Tan, Consultant, Principal Investigator — National Cancer Centre, Singapore
Locations (2):
- Singapore (2):
  - Singapore General Hospital, Singapore
  - National Cancer Centre Singapore, Singapore

REFERENCES:
- [Background] Lamberton GR, Hsi RS, Jin DH, Lindler TU, Jellison FC, Baldwin DD. Prospective comparison of four laparoscopic vessel ligation devices. J Endourol. 2008 Oct;22(10):2307-12. doi: 10.1089/end.2008.9715. PMID 18831673
- [Background] Harold KL, Pollinger H, Matthews BD, Kercher KW, Sing RF, Heniford BT. Comparison of ultrasonic energy, bipolar thermal energy, and vascular clips for the hemostasis of small-, medium-, and large-sized arteries. Surg Endosc. 2003 Aug;17(8):1228-30. doi: 10.1007/s00464-002-8833-7. Epub 2003 Jun 13. PMID 12799888
- [Background] Rahbari R, Mathur A, Kitano M, Guerrero M, Shen WT, Duh QY, Clark OH, Kebebew E. Prospective randomized trial of ligasure versus harmonic hemostasis technique in thyroidectomy. Ann Surg Oncol. 2011 Apr;18(4):1023-7. doi: 10.1245/s10434-010-1251-5. Epub 2010 Nov 12. PMID 21072688
- [Derived] Lee SH, Nguyen TK, Ong WS, Haaland B, Tay GC, Tan NC, Tan HK, Ng JCF, Iyer NG. Comparing the Utility and Surgical Outcomes of Harmonic Focus Ultrasonic Scalpel with Ligasure Small Jaw Bipolar Device in Thyroidectomies: A Prospective Randomized Controlled Trial. Ann Surg Oncol. 2019 Dec;26(13):4414-4422. doi: 10.1245/s10434-019-07806-w. Epub 2019 Sep 11. PMID 31512024